CLINICAL TRIAL: NCT00270985
Title: The Metabolic Effects of Almond Consumption in Adults With Pre-Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: Almond Board of California (Other)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0120050322
Record Dates: First submitted 2005-12-27; First posted 2005-12-29 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Prediabetes; Insulin Resistance; Metabolic Syndrome
Keywords: almonds; pre-diabetes; inflammatory; CRP
MeSH Terms: conditions — Prediabetic State; Insulin Resistance; Metabolic Syndrome; Glucose Intolerance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- nut free diet (Active Comparator): ADA recommended diabetes diet without any nuts
  Interventions: Behavioral: Nut free diet
- almond group (Experimental): calorie controlled diet with prescribed daily amount of almonds
  Interventions: Behavioral: Almonds in a calorie controlled diet

INTERVENTIONS:
Behavioral: Almonds in a calorie controlled diet — Prescribed daily dose of Almonds in calorie controlled diet for adults with pre-type 2 diabetes
  Arms: almond group
Behavioral: Nut free diet — Calorie controlled diet free of nuts for adults with pre-type 2 diabetes
  Arms: nut free diet

SUMMARY:
Study Hypothesis:

Daily consumption of almonds over 16 weeks will produce a decrease in hemoglobin A1c (HbA1c) levels in adults with pre-diabetes.

Lay Summary:

Persons developing type 2 diabetes mellitus (T2DM) will typically first have a condition called pre-diabetes. Lifestyle is a major factor that determines whether pre-diabetes becomes full T2DM. Lifestyle includes dietary habits and physical activity. Many people develop T2DM because of poor dietary habits and a sedentary lifestyle. Moreover, eating a high-fat, high-sugar diet can damage the blood vessels and increase the risk of strokes and heart attacks. A person's diet may produce substances in the blood that can interfere with the production of insulin in the pancreas. Sometimes, these changes in the insulin producing cells are serious and can eventually interfere with how the cells in the body use blood sugar, which causes T2DM. Techniques are available to measure circulating substances in the blood of persons with pre-diabetes that may be associated with the development of T2DM. Laboratory research has shown that almonds contain high levels of important compounds that may influence the onset of heart disease and T2DM. A meal plan that includes almonds daily will be given to half of the study participants and the other participants will be given a meal plan that is "nut-free". Because of the potential to delay the onset of heart disease and T2DM in some persons with pre-diabetes, this 16-week study will collect and analyze blood samples for changes that may make the person with pre-diabetes more likely to develop heart disease and T2DM. Blood samples will be collected at weeks 0, 8 and 16 to measure compounds that may be influenced by consuming almonds daily. This study will also attempt to understand other possible causes of heart disease and T2DM in persons with pre-diabetes; particularly those that might be related to body weight and body composition. Body composition techniques using very small amounts of electrical current are available to study body fat. Body weight, waist and hip measurements, blood pressure and body composition testing will be performed at the start of the study and every 4 weeks during the study. Lastly, these other possible causes of heart disease and T2DM will be investigated to look at relationships with the substances in the blood.

DETAILED DESCRIPTION:
Daily consumption of almonds over 16 weeks will produce a decrease in hemoglobin A1c (HbA1c) levels in adults with pre-diabetes.

Lay Summary:

Persons developing type 2 diabetes mellitus (T2DM) will typically first have a condition called pre-diabetes. Lifestyle is a major factor that determines whether pre-diabetes becomes full T2DM. Lifestyle includes dietary habits and physical activity. Many people develop T2DM because of poor dietary habits and a sedentary lifestyle. Moreover, eating a high-fat, high-sugar diet can damage the blood vessels and increase the risk of strokes and heart attacks. A person's diet may produce substances in the blood that can interfere with the production of insulin in the pancreas. Sometimes, these changes in the insulin producing cells are serious and can eventually interfere with how the cells in the body use blood sugar, which causes T2DM. Techniques are available to measure circulating substances in the blood of persons with pre-diabetes that may be associated with the development of T2DM. Laboratory research has shown that almonds contain high levels of important compounds that may influence the onset of heart disease and T2DM. A meal plan that includes almonds daily will be given to half of the study participants and the other participants will be given a meal plan that is "nut-free". Because of the potential to delay the onset of heart disease and T2DM in some persons with pre-diabetes, this 16-week study will collect and analyze blood samples for changes that may make the person with pre-diabetes more likely to develop heart disease and T2DM. Blood samples will be collected at weeks 0, 8 and 16 to measure compounds that may be influenced by consuming almonds daily. This study will also attempt to understand other possible causes of heart disease and T2DM in persons with pre-diabetes; particularly those that might be related to body weight and body composition. Body composition techniques using very small amounts of electrical current are available to study body fat. Body weight, waist and hip measurements, blood pressure and body composition testing will be performed at the start of the study and every 4 weeks during the study. Lastly, these other possible causes of heart disease and T2DM will be investigated to look at relationships with the substances in the blood.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* No self-reported allergy to almonds
* No history of irritable bowel disease or diverticulitis that could be exacerbated by daily almond intake
* Presence of pre-diabetes according to the 2005 American Diabetes Association diagnostic guidelines (fasting blood glucose between 100 to 125 mg/dl or casual blood glucose ≥ 140-199 mg/dl)
* Body mass index (BMI) 20-35 kg/m2 to enhance the generalizability of the study's findings to the population of adults with pre-diabetes
* Willingness to discontinue vitamin E supplement usage while enrolled in the study.

Exclusion Criteria:

* No concurrent use of corticosteroids or immunosuppressant medications (tacrolimus, cyclosporine, sirolimus, azathioprine, 6-mercaptopurine, mycophenolate mofetil, everolimus) in light of their effect on inflammatory biomarkers
* No liver disease, renal disease and/or severe dyslipidemia (triglycerides [TG] > 400mg/dl or total cholesterol [TC] > 300 mg/dl)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2006-01; Primary Completion 2007-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
HbA1c | 16 weeks
  change in HbA1c over the course of 16 wk intervention as an indication of blood glucose control

SECONDARY OUTCOMES:
hs-CRP | 16 wks
  change in high sensitivity C Reactive Protein as an indication of inflammation over course of the intervention
Il-6 | 16 weeks
  Change in Interleukin 6 over the 16 week intervention as an indication of inflammation/metabolic syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Gould Fogerite, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- UMDNJ, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available.

REFERENCES:
- [Result] Wien M, Bleich D, Raghuwanshi M, Gould-Forgerite S, Gomes J, Monahan-Couch L, Oda K. Almond consumption and cardiovascular risk factors in adults with prediabetes. J Am Coll Nutr. 2010 Jun;29(3):189-97. doi: 10.1080/07315724.2010.10719833. PMID 20833991